CLINICAL TRIAL: NCT00154050
Title: High Dose Candesartan Versus Quinapril for Restenosis Prophylaxis After Stent Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IKPD KARDCHEM 02-04
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Arterial Occlusive Diseases
Keywords: restenosis; intima hyperproliferation; stent angioplasty; pain-free walking distance
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — candesartan; Pharmaceutical Preparations; Quinapril

INTERVENTIONS:
Drug: candesartan (drug) or quinapril (drug)

SUMMARY:
The study is designed to test the hypothesis that high dose candesartan treatment compared to quinapril is able to reduce intima hyperproliferation and the restenosis rate after stent angioplasty in peripheral occlusive artery disease.

DETAILED DESCRIPTION:
Patients are randomly assigned to treatment with either candesartan 32 mg/d or Quinapril 20 mg/d before the angioplasty. Walking distance, intima media thickness and crurobrachial pressure ratios are compared after 6 weeks, 3 months and 6 months. After 6 months an angiographic control is performed.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* peripheral occlusive arterial disease Stad IIb Fontaine classification

Exclusion Criteria:

* patients with lesions not available for PTA
* renal insufficiency
* patients on calcium-antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2004-05; Study Completion 2006-07

PRIMARY OUTCOMES:
Restenosis/reintervention after 6 months

SECONDARY OUTCOMES:
pain-free walking distance
crurobrachial pressure ratios

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Chemnitz Hospital, Dept. of Internal Medicine I, Chemnitz, Germany